CLINICAL TRIAL: NCT02988024
Title: A Randomized, Open-Label, Single-Dose Study to Assess the Relative Bioavailability of LY03005 Oral Tablets Versus Pristiq Oral Tablets Under Fasting Conditions in Healthy Subjects
Brief Title: Pilot BA Study of New LY03005 vs Pristiq
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03005/CT-USA-103
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY03005 (Experimental): LY03005 80 mg
  Interventions: Drug: LY03005
- Pristiq (Active Comparator): Pristiq 50 mg
  Interventions: Drug: Pristiq

INTERVENTIONS:
Drug: LY03005 — LY03005
  Arms: LY03005
Drug: Pristiq
  Other Names: Desvenlafaxine
  Arms: Pristiq

SUMMARY:
The objects of this study is to assess the relative bioavailability (BA) of 80 mg LY03005 oral tablets compared to 50 mg Pristiq® oral tablets after a single oral intake under fasting conditions in healthy subjects between 18 and 50 years of age.

DETAILED DESCRIPTION:
Twenty (20) eligible subjects will be enrolled and assigned to either LY03005 group or Pristiq group at a 1:1 ratio at one site in the USA.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Male and female subjects between the ages of 18 and 50 years;
3. Considered healthy by the Principal Investigator, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
4. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening based on subject report;
5. Body mass index (BMI) of 19 to 30 kg/m 2 inclusive and body weight not less than 50 kg;
6. Willing and able to adhere to study restrictions and to be confined at the clinical research center.
7. All female subjects no matter of age must have a negative pregnancy test result at screening. In addition, female subjects must meet one of the following three conditions: (i) postmenopausal for at least 2 years, (ii) surgically sterile based on subject report, or (iii) if child-bearing potential, practicing or agree to practice an effective method of birth control by using an acceptable method of contraception.

Acceptable methods of birth control include oral, injected, vaginal or patch contraceptive, IUD (Intrauterine device)(copper intrauterine device), or double- barrier method (e.g., condom, diaphragm or cervical cap with spermicidal foam, cream, gel or suppository). Acceptable methods of birth control must be used for at least 14 days prior to the use of study drug, during the study and within one month after the end of the study.

Exclusion Criteria:

1. Clinically significant past history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, ophthalmological, or drug hypersensitivity;
2. History of suicide attempt in the past 12 months and/or seen by the investigators having a significant history of risk of suicide or homicide;
3. History or presence of malignancy other than adequately treated basal cell skin cancer;
4. Clinically relevant illness within one month prior to the screening visit or at screening visit that may interfere with the conduct of this study;
5. Subjects with a mean systolic blood pressure of three measurements >140 mmHg, or a mean diastolic blood pressure of three measurements >90 mmHg at screening;
6. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody;
7. A history of seizure. However, a history of febrile seizure is allowed;
8. A hospital admission or major surgery within 30 days prior to screening;
9. Participation in any other investigational drug trial within 30 days prior to screening;
10. A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
11. A history of alcohol abuse according to medical history within 6 months prior to screening;
12. A positive screen for alcohol, drugs of abuse;
13. Tobacco use within 6 months prior to screening based on subject report;
14. Subjects with hypersensitivity to PRISTIQ or medicines containing desvenlafaxine or its precursor venlafaxine;
15. Subjects who have participated in a previous clinical study of either LY03005 or PRISTIQ or medicines containing desvenlafaxine or its precursor, venlafaxine within 30 days prior to screening;
16. An unwillingness or inability to comply with food and beverage restrictions during study participation;
17. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
18. Use of prescription or over-the-counter (OTC) medications, and herbal (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) for the Pharmacokinetics (PK) of LY03005 | 4 days
  PK Samples drawn at 0 (within 30 minutes prior to dosing), 1,2,3,4 (+/- 5 min), 6,8,10,12,23,32,48 and 72 hours (+/- 15 min) after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Li, M.D., Study Chair — Luye Pharma Group Ltd.
Locations (1):
- Clinilabs, Inc., Eatontown, New Jersey, United States